CLINICAL TRIAL: NCT02377076
Title: Dietary Calcium Supplementation, Gut Permeability and Microbiota in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Dr Junia Maria Geraldo Gomes, Dr, Federal University of Vicosa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 526.005
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAIRY (Experimental): Dietary calcium supplementation
  Interventions: Dietary Supplement: Dietary calcium supplementation
- CONTROL (Placebo Comparator): Control
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Dietary calcium supplementation — Dietary calcium supplementation as milk powder
  Arms: DAIRY
Dietary Supplement: Control — Control (Whey protein, vitamin D, sugar and salt)
  Arms: CONTROL

SUMMARY:
Dietary calcium seems to act on glycemic control, favoring the prevention and treatment of type 2 diabetes mellitus (DM2). It is possible that calcium modulates gut microbiota and increase the integrity of the intestinal mucosa. This study aims to evaluate the effects of dietary calcium supplementation in permeability and intestinal microbiota in overweight type 2 diabetics. This is a single-blind, randomized, placebo-controlled, crossover study. Patients (n=20) with low habitual calcium intake will be allocated in control group (CONTROL) or test group (DAIRY). Hypocaloric diets (restriction of 500 kcal / day) will be prescribed containing 800 mg of calcium from dietary sources / day. During intervention period, a beverage (shake) (CONTROL - without the addition of calcium sources or DAIRY - 700 mg of calcium as milk powder) will be ingested in the laboratory. Food intake, body composition (total body fat and fat free mass) and anthropometric measures (waist circumference, waist-hip ratio, waist-height, neck circumference and sagittal abdominal diameter) will be evaluated at baseline and at the 6th and 12th weeks. Physical activity level, gut permeability, gut microbiota, and biochemical parameters (parathyroid hormone, 25-dihydroxy vitamin D, calcium, fasting glucose, fasting insulin, fructosamine, hemoglobin, HbA1c, uric acid, triglycerides, cholesterol total and partial, lipopolysaccharide, inflammatory markers) will be evaluated at baseline and after 12 weeks. The statistical analysis will be performed with the use of SPSS software (SPSS Inc., Chicago, IL, 2008, version 17.0). Parametric or non-parametric tests will be applied, according to the distribution of variables (level of statistical significance of 5%).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus using oral hypoglycemic medication
* Overweight (body mass index between 25 and 34.9 kg / m2)
* Usual intake of calcium less than 600 mg / day
* Level of physical activity light to moderate
* HbA1c above 7% or fasting glucose above 130 mg / dl

Exclusion Criteria:

* Smoking
* Use of calcium, vitamin D, magnesium, zinc, chromium, copper supplements or medication affecting the metabolism of these micronutrients,
* Use of drugs, herbs or diets that reduce appetite and body weight
* Estrogen replacement
* Gain or loss of at least 5 kg in the last 3 months
* Recent change in the level of physical activity
* Aversion or intolerance to food provided in the study
* Alcohol consumption of more than 2 doses / day (more than 50g ethanol / day)
* Eating disorders
* Endocrine disease, renal disease, hepatic disease or malabsorption syndrome that alters calcium metabolism
* History of recurrent nephrolithiasis
* Caffeine consumption of> 300 mg / day
* Pregnancy, lactation or postmenopausal
* Anemia
* Cardiovascular, infectious, inflammatory, thyroid, liver, kidney or intestinal disease
* Use of anti-inflammatory, antacids, antibiotics and laxatives drugs
* Major gastrointestinal surgery.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolism and body composition laboratory, Federal University of Vicosa, Viçosa, Minas Gerais, Brazil

REFERENCES:
- [Derived] Oliveira JSE, Gomes JMG, Costa JA, Oliveira LL, Alfenas RCG. Increased calcium intake from skimmed milk in energy-restricted diets reduces glycation markers in adults with type 2 diabetes and overweight: A secondary analysis of a randomized clinical trial. Nutr Res. 2024 Jul;127:40-52. doi: 10.1016/j.nutres.2024.04.008. Epub 2024 May 2. PMID 38861793
- [Derived] Gomes JMG, Costa JDA, Alfenas RCG. Effect of increased calcium consumption from fat-free milk in an energy-restricted diet on the metabolic syndrome and cardiometabolic outcomes in adults with type 2 diabetes mellitus: a randomised cross-over clinical trial. Br J Nutr. 2018 Feb;119(4):422-430. doi: 10.1017/S0007114517003956. PMID 29498351